CLINICAL TRIAL: NCT04370405
Title: A Phase 2, Single Arm, Open Label Clinical Study to Assess the Safety and Efficacy of YY-20394 in Subjects With Relapsed/Refractory Follicular Non-Hodgkin's Lymphoma
Brief Title: A Study of YY-20394 in Participants With Relapsed/Refractory Follicular Non-Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai YingLi Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YY-20394-002
Record Dates: First submitted 2020-04-28; First posted 2020-04-30 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Lymphoma, Follicular
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YY-20394 (Experimental): YY-20394 tablets will be given daily for 28 days in 28-day cycles until there appears evidence of progressive disease, intolerable toxicity, or the subject discontinues from the study treatment for other reasons.
  Interventions: Drug: YY-20394

INTERVENTIONS:
Drug: YY-20394 — YY-20394 tablets will be given daily for 28 days in 28-day cycles until there appears evidence of progressive disease, intolerable toxicity, or the subject discontinues from the study treatment for other reasons.

SUMMARY:
This is a study designed to evaluate the efficacy and safety of oral YY-20394 in patients with R/R follicular non-Hodgkin's lymphoma who have failed at least two prior systemic therapies.

DETAILED DESCRIPTION:
The study will be conducted in China to provide safety and efficacy data from this region. A Safety Run-in will be conducted to confirm the safety of the recommended Phase 2 dose (RP2D), 80 mg once daily, in a Asian population. PK samplings at Cycle 1, Day 1 will be taken.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥18 years of age at the time of signing the informed consent.
2. Has histologically or cytologically confirmed follicular non-Hodgkin's lymphoma
3. Has received at least two prior lines of systemic therapy (excluding radiation) for follicular lymphoma.(Has been treated with CD20 mAb and at least one alkylating agent, including but not limited to bendamostine, cyclophosphamide, isocyclophosphamide, chlorophenyl butylamine, Malan, busulfan, nitroso
4. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
5. Has a life expectancy >3 months.
6. Has radiographically measurable disease as per IRWG Criteria with at least one nodal lesion.
7. Fine organ function ANC≥1.0×109/L； PLT≥70×109/L(≥50×109/L in patients with bone marrow infiltration )； Hb≥80 g/L(≥70 g/L in patients with bone marrow infiltration)； TBIL≤1.5×ULN； Both ALT and AST≤2.5×ULN； Both BUN/Urea andCr≤1.5×ULN； LVEF≥50%； QTcF(QT interval corrected by friderica)Male<450 ms、Female<470 ms。
8. The washout period lasted at least four weeks of previous anti-tumor treatment (including radiotherapy, chemotherapy, hormone therapy, surgery or molecular targeted treatment) taken by the patient before the study to ensure complete clearance from the body.
9. Has adequate organ function as defined in Table 5 1. Specimen for this assessment must be collected within 14 days prior to the first dose of study treatment:
10. According to the judgment of the researchers, the patients can comply with the trial plan
11. The patient did not participate in the clinical trial as a subject within 1 month before the trial;

Exclusion Criteria:

* 1) Disease progress in the use of PI3kδ inhibitors 2) Pathological transformation of follicular non-Hodgkin's lymphoma to diffuse large B cell lymphoma 3) Any anti-tumor treatment within 4weeks. 4) Pathological fluid accumulations(such as hydrothorax and ascites )can not be controlled by drainage and other method in the third space 5) The dosage of steroid hormone (prednisone equivalent) was more than 20mg / day, and it was used continuously for more than 14 days 6) Has inability to swallow\ chronic diarrhea\ intestine obstruction snd other reasons that could have effluence on the administration and absorbtion. of the drug 7) Can't discontinue use of drugs (such as antiarrhythmic drugs) that may cause QT prolongation during the study.

  8) Lymphoma Patients with involvement of central nerve system. 9) Allergic constitution or known allergic history to the components of the drug.

  10) Has active effection of viruses\bacterium\ fungi and need to be treated(such as pneumonia ).

  11) Uncontrolled diabetes, pulmonary fibrosis, acute lung disease, interstitial lung disease, or liver failure 12) Has infection of HBV or HCV(Definition: HbsAg and/or HbcAb positive and the copy number of HBV DNA≥1×104/ml or ≥2000 IU/ml ) HCV antibody positive(acute or chornic effected actively) 13) Has history of immunodeficiency disease,include HIV positive or other acquired \ congenital immunodeficiency disease or history of allogeneic bone marrow organ transplangtation or history of hematopoietic stem cell transplangtation 14) Has received hematopoietic stem cell transplangtation within 90 days before the first dose of study treatment.

  15) Has any cardiac disease,including:(1)angina;(2) arrhythmias need to be clinical intervented;(3)myocardial infarction;(4)heart failure;(5)any other cardiac diseases that is not suitable for this trail according to the judgement of recheachers.

  16) Pregnant and lactating women or fertile women who have a positive pregnancy test 17) Has accompany diseases which do harm to the safety of patients or have impact on the study(such as server hypertension\diabetes\thyroid diseases ) 18) Has other kinds of malignant tumors except skin basal cell carcinoma and cervical carcinoma in situ

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Estimated)
Dates: Start 2019-04-29 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2021-02-22 (Estimated)

PRIMARY OUTCOMES:
Overall response rate, ORR | Throughout the study for approximately 2 years
  Overall response rate (ORRProportion of patients whose tumor volume reduces to a predetermined value and can maintain the minimum time limit-) assessed by an Independent Review Committee (IRC).

SECONDARY OUTCOMES:
Overall response rate (ORR) | Throughout the study for approximately 2 years
  Overall response rate (ORR-Proportion of patients whose tumor volume reduces to a predetermined value and can maintain the minimum time limit) assessed by reseachers.
Progression free survival, PFS | Throughout the study for approximately 2 years
  PFS, defined as the time from the first dose of study treatment to first documented disease progression or death due to any cause, whichever occurs first.
Overall survival, OS | Throughout the study for approximately 2 years
  The time from randomization to death for any reason.
Disease control rate, DCR | Throughout the study for approximately 2 years
  The percentage of cases with remission (PR+CR)and stable lesions(SD) after treatment in the number of evaluable cases.

CONTACTS AND LOCATIONS:
Locations (1):
- Hematology Hospital of Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China